CLINICAL TRIAL: NCT01187290
Title: Preoperative Chemoradiotherapy vs. Chemotherapy Alone in Nonsmall Cell Lung Cancer (NSCLC) Patients With Mediastinal Lymph Node Metastases (Stage IIIA, N2): A Randomized Prospective Phase II Trial
Brief Title: Preoperative Chemoradiotherapy Versus Chemotherapy Alone in Nonsmall Cell Lung Cancer (NSCLC) Patients With Mediastinal Lymph Node Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Luo qinquan, shanghai chest hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: chest1001
Record Dates: First submitted 2010-08-19; First posted 2010-08-24 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Preoperative chemoradiotherapy; stage IIIA, N2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neoadjuvant chemotherapy (No Intervention): Chemotherapy Docetaxel 75 mg/m2 1 hour iv infusion d1 Cisplatin 100 mg/m2 1 hour iv infusion d1 Schedule: 3 cycles repeated every 21 days
  Interventions: Radiation: neoadjuvant chemoradiotherapy
- neoadjuvant chemoradiotherapy (Experimental): Docetaxel 75 mg/m2 1 hour iv infusion d1 Cisplatin 100 mg/m2 1 hour iv infusion d1 Schedule: 3 cycles repeated every 21 days
  Interventions: Radiation: neoadjuvant chemoradiotherapy

INTERVENTIONS:
Radiation: neoadjuvant chemoradiotherapy — Radiotherapy (3 weeks after last chemotherapy administration) 44 Gy in 22 fractions concomitant boost technique in 3 weeks

SUMMARY:
The main objective of this trial is to compare feasibility and efficacy of sequential neoadjuvant chemoradiotherapy with 44Gy concomitant boost to neoadjuvant chemotherapy alone. Secondary objectives are to assess the value of position emission tomography (PET）in predicting pathological response and event-free survival（EFS）in stage IIIA non-small cell lung cancer (NSCLC). Further to compare the amount of serum DNA in patients with stage IIIa NSCLC before, during and after chemotherapy, before and after radiotherapy (in arm A) and during follow-up in patients randomized into the trial and to correlate the Deoxyribonucleic acid (DNA) variation with tumor response, remission duration and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NSCLC with nodal metastases: T1-3N2M0
* Performance status 0-1
* Patient medically fit enough for protocol therapy, including operability
* Age 18-75
* Written informed consent
* No previous chemo- or radiotherapy

Exclusion Criteria:

* Patients with prior or concomitant malignancies Allowed are: non-melanomatous skin cancer, adequately treated in situ cervical cancer or any other neoplastic diseases with disease-free interval ³ 5 years.
* Presence or history of any distant metastasis
* Unstable cardiac disease requiring treatment, congestive heart failure or angina pectoris even if medically controlled, significant arrhythmia, or prior history of myocardial infarction in the last 3 months
* History of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
* Active uncontrolled infection
* Uncontrolled diabetes mellitus
* Gastric ulcers
* Preexisting peripheral neuropathy (> grade 1)
* Other serious underlying medical condition which could impair the ability of the patient to participate in the trial
* Concurrent treatment with other experimental drugs
* Pretreatment with any other cytostatic therapy
* Previous radiotherapy to the chest
* Concurrent treatment with prednisone (or equivalent) except: for the prophylactic medication regimen before treatment, treatment of acute hypersensitivity reactions or chronic treatment (initiated > 6 months prior to trial entry) at low dose (£ 20 mg methylprednisolone or equivalent)
* Definite contraindications for the use of corticosteroids as premedication
* Treatment within a clinical trial within 30 days prior to trial entry
* Socioeconomic or geographic circumstances that may prohibit proper staging, treatment or follow-up procedures
* Pregnancy, lactation period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | five years

SECONDARY OUTCOMES:
Operability | within the first 30 days (plus or minus 3 days) after surgery
Postoperative 30-day mortality | 30 days after treatment
Toxicity | 30 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: luo qingquan, M.D., Study Chair — Shanghai Chest Hospital